CLINICAL TRIAL: NCT06681935
Title: Defining Mechanisms of Surgical Site Infection After Oral Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Joseph Zenga, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO00052346; R21DE032844 (NIH)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Oral Cancer
Keywords: Surgical Site Infection; Oral Cavity Reconstruction
MeSH Terms: conditions — Mouth Neoplasms; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole genome sequencing may be included as part of the genetic testing for this research. Genetic testing will only be performed on microbial samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects undergoing Oral Cavity Reconstruction: The cohort will be oral cancer patients undergoing standard of care oral cavity reconstruction.
  Interventions: Procedure: Oral Cavity Reconstruction

INTERVENTIONS:
Procedure: Oral Cavity Reconstruction — This procedure includes a planned surgical connection from the oral cavity to the neck soft tissues which is repaired through free or pedicled flap reconstruction.

SUMMARY:
The study design is an observational cohort study of patients undergoing standard of care oral cavity reconstruction. An observational study is required to prospectively evaluate microbial and antibiotic mechanisms underlying surgical site infection after oral cavity reconstruction.

DETAILED DESCRIPTION:
This is a single institution study at the Medical College of Wisconsin, given the feasibility of projected sample size accrual as well as the clinical and translational expertise at this location for investigating surgical site infection after oral cavity reconstruction. Biospecimens collected will include oral, nasal, pharyngoesophageal, and skin microbial swabs, blood, and discard tissue samples obtained during standard of care oral cavity reconstruction surgery and an oral swab and nasal swab obtained post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed and dated informed consent form. Subjects must have the capacity to consent for themselves.
2. Willing to comply with all study procedures and be available for the duration of the study.
3. Aged 21 years or older.
4. Planned to undergo standard of care oral cavity reconstruction surgery with use of ampicillin/sulbactam as the prophylactic antibiotic agent administered.
5. Oral cavity reconstruction surgery will be defined as any surgical procedure which includes a planned connection from the oral cavity to the neck soft tissues which is repaired with a free or regional tissue flap.
6. History of oral or oropharyngeal cancer.

Exclusion Criteria:

1. Allergy to ampicillin/sulbactam.
2. Vulnerable populations including pregnant women and prisoners.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The projected sample size is 40 patients over 2 years. The cohort will be oral cancer patients undergoing standard of care oral cavity reconstruction, which includes a planned surgical connection from the oral cavity to the neck soft tissues which is repaired through free or pedicled flap reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Source of bacteria leading to a surgical site infection | Up to 30 days
  This is the number of subjects with surgical site infections with bacteria that originates from the oral cavity. This will be determined by metagenomic mapping of bacterial strains causing surgical site infection back on to the metagenomic samples from their anatomic source (oral cavity, nasal cavity, pharyngoesophagus, donor site skin).

SECONDARY OUTCOMES:
Tissue antibiotic correlations | Up to 30 days
  This is the number of subjects with tissue antibiotic concentrations that correlate with surgical site infection. This will be accomplished by liquid chromatography/mass spectrometry (LC-MS) to assess for antibiotic concentration in tissue and blood during surgery.
Plasma antibiotic correlations | Up to 30 days
  This is the number of subjects with plasma antibiotic concentrations that correlate with surgical site infection. This will be accomplished by liquid chromatography/mass spectrometry (LC-MS) to assess for antibiotic concentration in tissue and blood during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zenga, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No